CLINICAL TRIAL: NCT00748163
Title: Phase II Study of ABI-007 Plus Sunitinib as First Line Treatment for Non-Small Cell Lung Cancer
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation and Sunitinib as First-Line Therapy in Treating Patients With Stage IV Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been abandoned for lack of available funding.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007LS098; 0802M26201 (Other: IRB, University of Minnesota); ABX080 (Other: Abraxis); GA6181W (Other: Pfizer)
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Lung Cancer
Keywords: stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Taxes; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stage IV Non-Small Cell Lung Cancer Patients (Experimental): Patients with stage IV non-small cell lung cancer treated with paclitaxel albumin-stabilized nanoparticle formulation and sunitinib malate as first-line therapy.
  Interventions: Drug: paclitaxel albumin-stabilized nanoparticle formulation; Drug: sunitinib malate

INTERVENTIONS:
Drug: paclitaxel albumin-stabilized nanoparticle formulation
Drug: sunitinib malate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving paclitaxel albumin-stabilized nanoparticle formulation together with sunitinib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel albumin-stabilized nanoparticle formulation together with sunitinib works as first-line therapy in treating patients with stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the tumor response rate in patients with stage IV non-small cell lung cancer treated with paclitaxel albumin-stabilized nanoparticle formulation and sunitinib malate as first-line therapy.

Secondary

* To determine the time to objective tumor response and duration of response in responding patients.
* To determine the time to treatment failure and overall survival of these patients.
* To characterize the toxicities of this regimen in these patients.

OUTLINE: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Patients also receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 8 weeks until disease progression and then every 3 months for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IV disease
* At least 1 measurable lesion as defined by modified RECIST criteria
* No symptomatic or untreated brain metastases

  * Prior brain metastases allowed provided the CNS disease has been treated and is considered stable and the patient has recovered from the acute toxic effects of the treatment prior to study entry

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-1
* WBC ≥ 3.0 x 10^9/L
* ANC ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (≤ 5 times ULN if liver has tumor involvement)
* Creatinine ≤ 1.5 mg/dL
* LVEF ≥ 40% by MUGA
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment

Exclusion criteria:

* Congestive heart failure, myocardial infarction, or coronary artery bypass graft within the past 12 months
* Ongoing severe or unstable angina
* Unstable arrhythmia requiring medication
* Sensory neuropathy ≥ grade 2 (according to NCI CTCAE v3.0)
* Known hypersensitivity to any of the agents used in this study
* Serious medical or psychiatric illness that, in the opinion of the enrolling investigator, is likely to interfere with study participation

PRIOR CONCURRENT THERAPY:

* No prior systemic therapy for NSCLC
* More than 4 weeks since prior major surgery
* More than 7 days since prior and no concurrent potent CYP3A4 inhibitors, including any of the following:

  * Ketoconazole
  * Itraconazole
  * Clarithromycin
  * Erythromycin
  * Diltiazem
  * Verapamil
  * Delavirdine
  * Indinavir
  * Saquinavir
  * Ritonavir
  * Atazanavir
  * Nelfinavir
* More than 12 days since prior and no concurrent potent CYP3A4 inducers, including any of the following:

  * Rifampin
  * Rifabutin
  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * St. John's wort
  * Efavirenz
  * Tipranavir
* No concurrent treatment with a drug having proarrhythmic potential, including any of the following:

  * Terfenadine
  * Quinidine
  * Procainamide
  * Disopyramide
  * Sotalol
  * Probucol
  * Bepridil
  * Haloperidol
  * Risperidone
  * Indapamide
  * Flecainide
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08 (Estimated); Primary Completion 2008-08 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Response rate | 1 Year

SECONDARY OUTCOMES:
Time to objective tumor response as assessed by RECIST criteria | 1 Year
Duration of response | 1 Year
Time to treatment failure | 1 Year
Overall survival | 1 Year
Toxicity and adverse events as assessed by NCI CTCAE v3.0 | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Dudek, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota